CLINICAL TRIAL: NCT03582696
Title: Carolina Heart Alliance Networking for Greater Equity (CHANGE)
Brief Title: Carolina Heart Alliance Networking for Greater Equity
Acronym: CHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-2822; 5U48DP005017-04 (NIH)
Record Dates: First submitted 2018-06-19; First posted 2018-07-11 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Cardiovascular Disease (CVD)
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The participants who are engaged with CHWs will be assessed in terms of weight and blood pressure compared to pre-intervention levels and will also complete pre and post dietary and physical activity questionnaires.
Oversight: Data Monitoring Committee: No

ARMS (1):
- No Arms (Other): Participants are not assigned to randomized study arms or groups.
  Interventions: Behavioral: CHANGE Study

INTERVENTIONS:
Behavioral: CHANGE Study — The CHANGE strategy is designed to improve the dissemination and implementation of CVD EBIs by strengthening clinical-community linkages

SUMMARY:
In North Carolina, and nationally, cardiovascular disease (CVD) is the leading cause of death and disease among adults. North Carolina adults have high rates of CVD behavioral risk factors such as physical inactivity, unhealthy eating habits, smoking, and being overweight and obese. To help reduce these risks, researchers from the University of North Carolina at Chapel Hill Prevention Research Center (UNC PRC) will test the effectiveness and implementation of Carolina Heart Alliance Networking for Greater Equality (CHANGE).

CHANGE is a health promotion strategy to link public health and clinical services through community health workers (CHWs). Primary care clinics, public health, and CHWs all have strengths in addressing chronic disease risk factors, but there is a widely recognized gap in the coordination among them. The CHANGE strategy will use CHWs as members of primary care and public health teams to distribute a behavioral change intervention called Heart-to-Health to a total of 480 clinic patients at risk for CVD. Heart-to-Health is an effective lifestyle and medication adherence intervention that includes a computerized decision aid to guide delivery of tailored counseling sessions. The counseling sessions are focused on diet, physical activity, tobacco cessation, and medication adherence and are facilitated by CHWs using tablet computers. The CHWs will use tablet computers to communicate with a medical home team about important patient health information to be acted on in real time. The CHWs also will link participants to public health and other community based resources to support behavior change. The CHANGE strategy will be tested in one underserved, rural community and then replicated in a second community.

Researchers from the UNC PRC will examine whether CHANGE is effective at increasing the reach of clinic and public community services to at risk populations and at improving composite coronary heart disease risk.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of mortality and morbidity among North Carolina (NC) and US adults, yet evidence-based CVD prevention interventions are often minimally implemented and poorly integrated across community and clinical settings. To address this gap, we will develop and test a multi-component strategy to help communities effectively implement evidence-based interventions (EBIs) to prevent CVD. We call our strategy the Carolina Heart Alliance Networking for Greater Equity (CHANGE) strategy. The CHANGE strategy will specifically address NC's large underserved, rural population, which is at increased risk for CVD due in part to behavioral risk factors, including physical inactivity, poor diet, and tobacco use.

The CHANGE strategy is designed to improve the dissemination and implementation of CVD EBIs by strengthening clinical-community linkages. Clinics have strengths in identifying individuals at high risk for cardiovascular disease and prescribing medications and behavioral change to mitigate risk. However, clinics only reach those who seek care, and most clinics lack the capacity to deliver behavioral change EBIs. Public health has strengths in implementing behavioral and environmental change EBIs in the communities where people live. Therefore, the core focus of the CHANGE strategy is to create new structures to leverage the complementary strengths of clinics and public health departments, thereby expanding the reach and effectiveness of both clinic- and community-based EBIs. Because of their potential to reach underserved populations, community health workers (CHWs) are at the center of the CHANGE strategy. Working as part of a clinic/public health collaboration, CHWs will deliver a behavioral change EBI (Heart-to-Health). By linking and leveraging clinical and public health prevention activities, new opportunities for individuals and communities to reduce their risk for CVD will be created. CHWs will be equipped with tablet computers that provide decision support for delivering Heart-to-Health and facilitate linkages among clinics, public health, and community services. Linking services within complex systems is challenging, and many good ideas fall short at the level of implementation. Therefore, the study will apply an effectiveness-implementation hybrid design with a primary focus on the effective implementation of the CHANGE strategy and a secondary focus on its effectiveness at reducing CVD risk. With support and input from community stakeholders the investigators will refine the CHANGE strategy (Year 1), test it in one underserved, rural community (Years 2-3) and then replicate it in a second community (Years 4-5).

Guided by key constructs from implementation science53 and the expanded Chronic Disease Model,54 the study's specific aims are as follows:

Aim 1. Refine the CHANGE strategy through community-engaged formative research to:

(a) identify existing CVD-related clinic and community services and barriers to their use, (b) engage stakeholders in designing the CHWs' roles and systems for integrating their work within clinical and public health practice, and (c) assess the tablet's usability for decision-support and data transfer.

Aim 2. Assess the CHANGE strategy's implementation and effectiveness. Aim 2a. Use an explanatory sequential mixed-methods approach55 to assess the strategy's

(1) Best processes for engaging partners and building capacity to plan and implement EBIs. (2) Effectiveness at increasing the reach of CVD-related public health EBIs.56 (3) Other Implementation outcomes (fidelity, cost, sustainability, acceptability, and feasibility).53

Aim 2b. Use a pre-post comparison design to confirm the effectiveness of Heart-to-Health at improving composite coronary heart disease risk (primary outcome = Framingham Risk Score) and related risk factors: blood pressure, blood lipids, diet quality, physical activity, and tobacco use.

Aim 2c. Use a matched control, pre-post comparison design to assess the overall CHANGE strategy's effects on the proportion of the clinic's total at-risk population that have cholesterol and blood pressure under control as compared to three matched comparison clinics.

Aim 3. Plan for taking the CHANGE strategy to scale by replicating it in one additional community, identifying its core components,57, 58 creating and disseminating a replication toolkit, and promoting the strategy's adoption through NC's multiple clinical, public health, and research networks.

The CHANGE Project seeks to recruit 380 adults who live or receive health care in Hertford County (Phase I) or Edgecombe/Nash Counties (Phase II) and are at risk of CVD. The investigators have completed enrollment in Herford County and are about to begin enrollment in Edgecombe/Nash. Through a series of 4 in-person and 3 phone sessions, 2 CHWs will meet with adults who are at risk of CVD to provide health information, support in setting behavioral goals and referrals to community resources. The CHWs' intervention activities are adapted from the evidence-based Heart-to-Health curriculum for individual behavior change. Outcomes will be measured using pre- post- data from all enrolled participants, including pre- post- CVD risk score (Framingham Risk Score (FRS) or the atherosclerotic cardiovascular disease (ASCVD)) data from a participant subgroup. Process outcomes will be assessed using a tracking tool designed specifically for this study to facilitate the CHWs' data collection, intervention delivery, and case management activities in the field. Interviews will be conducted with program participants within a month of the final study visit to better understand their experience with the CHANGE program.

ELIGIBILITY:
Inclusion Criteria:

* Participants are adults ages 18-80 years old who are residents of Hertford, Edgecombe or Nash County, North Carolina or receive public health or healthcare services in Hertford, Edgecombe or Nash County, NC. Additionally, subjects enrolled and receiving services from Roanoke Chowan Community Health Center and OIC Family Medicine AND at elevated risk of a cardiac event. Individuals are at elevated risk if they are represented in any of the following five groups of clinic patients:

Group 1: ages 18-80. With no diabetes and no CVD. And, with high blood pressure (HBP) and high cholesterol;

Group 2: ages 65-80. With no diabetes and no CVD. And, with HBP or high cholesterol;

Group 3: ages 18-80. With diabetes and no CVD. And, with one or more of the following risk factors: HBP, high cholesterol and/or elevated average blood glucose measure;

Group 4: 55-64. With CVD. And, with two or more of the following risk factors: HBP, high cholesterol and/or elevated average blood glucose measure;

Group 5: 65-80. With CVD. And, with one or more of the following: HBP, high cholesterol and/or elevated average blood glucose measure.

Exclusion Criteria:

* Individuals who do not speak English will be excluded from the study because our intervention materials and activities will not be translated into any other languages at this time. We will exclude or withdraw women who report that they are pregnant as pregnancy may account for any changes in weight, BMI and blood pressure.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2016-09-11 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Disease risk score change | 4 months
  Will use the ASCVD pooled 10-year risk calculation to determine estimated 10 year risk of heart attack stroke or death (range 0-100). Will reassess after the 4 month intervention.

SECONDARY OUTCOMES:
Weight | 4 months
  Compare pre-intervention with post-intervention weight
Systolic blood Pressure (SBP) | 4 months
  Compare pre-intervention SBP with post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Cykert, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - Roanoke Chowan Community Health Center, Ahoskie, North Carolina
  - OIC Family Medical Center, Rocky Mount, North Carolina
  - Edgecombe Health Department, Tarboro, North Carolina
  - Hertford County Public Health Authority, Winton, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samuel-Hodge CD, Ziya Gizlice, Allgood SD, Bunton AJ, Erskine A, Leeman J, Cykert S. A Hybrid Implementation-Effectiveness Study of a Community Health Worker-Delivered Intervention to Reduce Cardiovascular Disease Risk in a Rural, Underserved Non-Hispanic Black Population: The CHANGE Study. Am J Health Promot. 2022 Jul;36(6):948-958. doi: 10.1177/08901171221078272. Epub 2022 Apr 14. PMID 35422132
- [Derived] Samuel-Hodge CD, Gizlice Z, Allgood SD, Bunton AJ, Erskine A, Leeman J, Cykert S. Strengthening community-clinical linkages to reduce cardiovascular disease risk in rural NC: feasibility phase of the CHANGE study. BMC Public Health. 2020 Feb 21;20(1):264. doi: 10.1186/s12889-020-8223-x. PMID 32085707